CLINICAL TRIAL: NCT07379788
Title: Mitral Remodeling Index: A Novel Composite Measure the Effect of ARNI Alone Versus ARNI Combined With SGLT2 Inhibitors on Functional Mitral Regurgitation Remodeling.
Brief Title: ARNI Combined With SGLT2 Inhibitors on Functional Mitral Regurgitation Remodeling
Status: Recruiting | Type: Observational
Sponsor: Rehab Werida (Other)
Collaborators: Tanta University (Other); Madinah Cardiac Center in Madinah, KSA. (Unknown)
Responsible Party: Sponsor-Investigator, Rehab Werida, Associate Professor, Damanhour University
Organization: Damanhour University (Other)
Other Study IDs: ARNI, SGLT2 Inhibitors & MRI
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Left atrial volume index (LAVI); Mitral Remodeling Index (MRIx); left ventricular ejection fraction (LVEF); functional mitral regurgitation (FMR)
MeSH Terms: conditions — Heart Failure | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARNI Monotherapy Group:: Patients receiving sacubitril/valsartan without concomitant SGLT2 inhibitor therapy.
  Interventions: Drug: Sacubitril/Valsartan 49 MG-51 MG Oral Tablet [ENTRESTO]
- Combination Therapy Group:: Patients receiving sacubitril/valsartan in combination with an SGLT2 inhibitor (empagliflozin 10 mg daily).
  Interventions: Drug: Empagliflozin10Mg Tab

INTERVENTIONS:
Drug: Sacubitril/Valsartan 49 MG-51 MG Oral Tablet [ENTRESTO] — Patients receiving Sacubitril/Valsartan 49 MG-51 MG Oral Tablet without concomitant SGLT2 inhibitor therapy.
  Other Names: Entresto
  Groups: ARNI Monotherapy Group:
Drug: Empagliflozin10Mg Tab — Combination Therapy Group: Patients receiving Sacubitril/Valsartan 49 MG-51 MG Oral Tablet in combination with an SGLT2 inhibitor (empagliflozin 10 mg daily).
  Other Names: Empagliflozin10Mg plus Sacubitril/Valsartan 49 MG-51 MG Oral Tablet
  Groups: Combination Therapy Group:

SUMMARY:
This study aimed to compare the effects of ARNI monotherapy versus combined ARNI and SGLT2 inhibitor therapy on Mitral Remodeling Index (MRIx) and Functional mitral regurgitation (FMR) remodeling in patients with heart failure with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
This was a retrospective observational cohort study conducted at Madinah Cardiac Center (MCC), Saudi Arabia, a tertiary referral center with a high-volume heart-failure unit and advanced echocardiographic services. Consecutive patients with chronic heart failure with reduced ejection fraction (HFrEF) and functional mitral regurgitation (FMR) were enrolled between [January 2025] and [December 2025].

Eligible patients were on sacubitril/valsartan (ARNI), either as monotherapy or in combination with a sodium-glucose cotransporter-2 (SGLT2) inhibitor, according to contemporary heart failure guidelines and treating physician discretion.

The study protocol conformed to the principles of the Declaration of Helsinki and was approved by the local institutional ethics committee; Madinah Cardiac Center before the beginning of the study.

• Treatment Groups

Patients were stratified into two groups based on pharmacological therapy:

1. ARNI Monotherapy Group: Patients receiving sacubitril/valsartan without concomitant SGLT2 inhibitor therapy.
2. Combination Therapy Group: Patients receiving sacubitril/valsartan in combination with an SGLT2 inhibitor (empagliflozin 10 mg daily).

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* left ventricular ejection fraction (LVEF) <50%;
* Presence of functional mitral regurgitation (mild, moderate, or severe) on transthoracic echocardiography; and
* stable sinus rhythm or controlled atrial fibrillation.

Exclusion Criteria:

* primary (degenerative or rheumatic) mitral valve disease,
* prior mitral valve surgery or transcatheter intervention,
* acute decompensated heart failure within four weeks,
* significant primary valvular disease other than FMR,
* severe renal impairment (estimated glomerular filtration rate <30 mL/min/1.73 m²),
* inadequate echocardiographic image quality.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: • Treatment Groups
  Patients were stratified into two groups based on pharmacological therapy:
  1. ARNI Monotherapy Group: Patients receiving Sacubitril/Valsartan 49 MG-51 MG Oral Tablet without concomitant SGLT2 inhibitor therapy.
  2. Combination Therapy Group: Patients receiving Sacubitril/Valsartan 49 MG-51 MG Oral Tablet sacubitril/valsartan in combination with an SGLT2 inhibitor (empagliflozin 10 mg daily).
  Sacubitril/valsartan was initiated and up titrated to the maximally tolerated dose according to guideline recommendations (13). SGLT2 inhibitors were prescribed at standard approved doses. Background heart failure therapy, including beta-blockers and mineralocorticoid receptor antagonists, was maintained whenever clinically feasible.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-12-25 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
LVEF % | 6 months
  Change in left ventricular ejection fraction percent
Left Atrial Volume index (LAVI) | 6 months
  Change Left Atrial Volume index (LAVI)
Mitral Remodeling Index | 6 months
  Change in Mitral Remodeling Index
Peak GLS number | 6 months
  Change in Peak Global Longitudinal Strain

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa Khedr, Ass Prof., Study Director — Madina Cardiac Center, KSA
Locations (1):
- Madinah Cardiac Center, Madinah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Verma S, McMurray JJV. SGLT2 inhibitors and mechanisms of cardiovascular benefit: a state-of-the-art review. Diabetologia. 2018 Oct;61(10):2108-2117. doi: 10.1007/s00125-018-4670-7. Epub 2018 Aug 22. PMID 30132036